CLINICAL TRIAL: NCT05148715
Title: Calcineurin Inhibitor in NEuRoloGically Deceased Donors to Decrease Kidney delaYed Graft Function (CINERGY)-Pilot Trial
Brief Title: Calcineurin Inhibitor in NEuRoloGically Deceased Donors to Decrease Kidney delaYed Graft Function (CINERGY)
Acronym: CINERGY
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP-31-2020-3348
Record Dates: First submitted 2021-10-18; First posted 2021-12-08 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Organ Transplant Failure or Rejection; Brain Death; Ischemic Reperfusion Injury
Keywords: organ donation and transplantation
MeSH Terms: conditions — Rejection, Psychology; Brain Death | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tacrolimus (Experimental): Tacrolimus 0.02 mg/kg ideal body weight 4-8 hours before organ recovery
  Interventions: Drug: Tacrolimus
- Placebo (Placebo Comparator): 0.9% sodium chloride 4-8 hours before organ recovery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tacrolimus — Single dose intravenous tacrolimus over 4 hour infusion at a dose of 0.02 mg/kg ideal body weight diluted with 0.9% sodium chloride starting 4-8 hours before scheduled organ recovery.
  Other Names: Prograf
  Arms: Tacrolimus
Drug: Placebo — Single dose of intravenous 0.9% sodium chloride over 4 hour infusion, starting 4-8 hours before scheduled organ recovery.
  Arms: Placebo

SUMMARY:
The investigators hypothesize that preconditioning neurologically deceased organ donors with the calcineurin inhibitor tacrolimus will improve short and long-term transplant survival without causing harm. Organ donors will be randomized to receive either 0.02 mg/kg ideal body weight (IBW) of tacrolimus single infusion or placebo before organ recovery. All corresponding recipients are enrolled and data is collected up to 7 days post-transplant to determine graft function and at 1 year to collect outcomes of vital status, re-transplantation and dialysis. The CINERGY Pilot Trial assesses feasibility for the main trial.

DETAILED DESCRIPTION:
Background: Organ donation saves lives, and improves quality of life for thousands of people. But organ donation falls short of expectations for some patients who suffer early graft loss. During organ donation surgery, the supply of blood with oxygen and nutrients is suspended. When restored during transplant surgery, a cascade of inflammation perturbs the newly transplanted organ -causing ischemia-reperfusion injury. When severe, it can hinder transplant function in the early post-operative period, lead to profound critical illness, increase the risks of transplant rejection and chronic disease, and reduce the transplant lifespan. Administration of tacrolimus, a calcineurin inhibitor, to neurologically deceased donors may reduce ischemia-reperfusion injury in transplant recipients.

Objectives: The CINERGY Pilot Trial will test the feasibility of comparing tacrolimus to placebo for the prevention of delayed graft function in kidney recipients and establish the foundation for a large, multi-centre randomized controlled trial (RCT).

Methods: 90 neurologically deceased kidney donors will be randomized to either tacrolimus (0.02 mg/kg) or the corresponding placebo 4-8 hours before organ recovery. To be included in the CINERGY Pilot RCT, donors will need to meet inclusion criteria. All corresponding recipients are enrolled and their data is collected in the first 7 days and at 12 months after transplantation.

Outcomes: Feasibility: Donor accrual rate and consent rate of organ recipients. Safety: acute kidney injury, hyperkalemia and anaphylaxis in donors and recipients. Clinical: graft function within 7 days in all recipients, vital status, re-transplantation and need for dialysis at 12 months.

Relevance: This pilot study will inform the feasibility and design of a larger trial. Moreover, the CINERGY Pilot RCT will pave the way for future trials linking organ donation and transplantation across Canada.

ELIGIBILITY:
Neurologically deceased donors who meet the inclusion and exclusion criteria will be eligible for participating in this study along with the correlating organ recipients who meet inclusion criteria.

Donor Inclusion Criteria:

* ≥18 years of age;
* Neurologically deceased;
* Consent for deceased organ donation;
* All organ recipients have been identified;
* ≥ 1 kidney allocated to a recipient.

Donor Exclusion Criteria:

* Known hypersensitivity to tacrolimus or polyoxyl 60 hydrogenated castor oil;
* One or more organs allocated to a non-participating transplant program;
* Unlikely access to study drug (e.g., due to supply issues, or pharmacist availability);
* One or more organ recipients has not agreed to receive an organ from a donor participating in the study;
* One or more organs are allocated to a recipient under the age of 18;
* A transplant physician has judged that donor tacrolimus will be unsuitable for an intended recipient.

Recipient Inclusion Criteria

* Organ/Transplant graft originated from a donor enrolled in this study.

No exclusion criteria.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Organ donor accrual rates | 6 to 12 months after the beginning of the trial
  One primary objective of this pilot study is to determine if a national multi-centre placebo randomized controlled trial (RCT) will be feasible with respect to: organ donor accrual.
Recipient consent rate | 6 to 12 months after the beginning of the trial
  Another primary objective of this pilot study is to determine if a national multi-centre placebo controlled RCT will be feasible with respect to the consent rates of organ recipients. Recipient consent rates will be assessed during analysis, analyzing the rate and reasons for non-enrolment.

SECONDARY OUTCOMES:
Correlation between two methods for obtaining survival status | 12 months post transplant
  We will compare 2 methods (Hospital records, Canadian Institute for Health Information) for obtaining recipient survival at 12 months post-transplant.
Unexpected adverse events | Within 7 days post transplant
  In donors and recipients, unexpected adverse events as identified by clinical staff will be reported and analyzed.
Percentage of donors with acute kidney injury (AKI) | Within 4 hours after the end of the study drug infusion
  AKI defined as defined as Kidney disease: Improving global outcome (KDIGO) stage II (or more): serum creatinine ≥ 2.0 times baseline OR a urine output <0.5mL/kg/h for ≥12 hours
Percentage of donors with hyperkalemia | Within 4 hours after the end of the study drug infusion
  Hyperkalemia defined as a potassium level > 5 mmol/L
Percentage of donors hypertension during tacrolimus infusion | Within 4 hours after the initiation of study drug infusion
  Hypertension (systolic blood pressure ≥ 160 mmHg or mean arterial pressure ≥ 90 mmHg for > 15 minutes)
Percentage of donors with cardiac arrhythmia associated with tacrolimus infusion | Within 4 hours after the initiation of study drug infusion
  Cardiac arrhythmias defined as new onset of atrial fibrillation or flutter, ventricular tachycardia or fibrillation
Percentage of donors with anaphylaxis | Within 4 hours after the initiation of study drug infusion
  Anaphylaxis defined as per The American Academy of Allergy, Asthma and Immunology
Percentage of recipients with acute kidney injury | Within 7 days post transplant
  AKI defined as defined as KDIGO stage II or more: serum creatinine ≥ 2.0 times baseline OR a urine output <0.5mL/kg/h for ≥12 hours
Percentage of recipients with hyperkalemia | Within 7 days post transplant
  Hyperkalemia defined as a potassium level > 5 mmol/L
Percentage of recipients with anaphylaxis | Within 7 days post transplant
  Anaphylaxis defined as per The American Academy of Allergy, Asthma and Immunology
Recipient serum tacrolimus levels | Within 7 days post transplant
  Clinical research staff will abstract routine serum tacrolimus levels (when measured) from hospital records over the first 7 days, along with local thresholds for toxic level.
Percentage of liver recipients with early graft function | Within 7 days post transplant
  At least ≥ 1 of the following criteria: Bilirubin ≥ 10 mg/dL , International normalized ratio (INR) ≥ 1.6 AST or ALT level > 2000 IU/
Graft survival | 12 months post transplant
  Need to be re-transplanted or to be on the re-transplant list.
Recipient survival | 12 months post transplant
  Recipient death
Recipients requiring dialysis | 12 months post transplant
  Recipient requirement for dialysis at 12 months
Percentage of lungs recipients with severe primary graft dysfunction | Within 3 days post transplant
  PaO2/FiO2 ratio <200 and diffuse infiltration/pulmonary edema on chest radiograph
Percentage of kidney recipients with delayed graft function | Within 7 days post transplant
  Requirement of ≥ 1 hemodialysis session
Percentage of heart recipients with severe primary graft dysfunction | Within 1 days post transplant
  Dependence on mechanical support
Percentage of pancreas recipients with delayed graft function | At hospital discharge, an average of 7 days
  Requirement of ≥1 exogenous insulin at hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Frédérick D'Aragon, Principal Investigator — Université de Sherbrooke; Maureen Meade, Principal Investigator — McMaster University; Markus Selzner, Principal Investigator — University of Toronto
Locations (9):
- Canada (9):
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - L'Institut de Cardiologie de Montréal, Montreal, Quebec
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre Hospitalier Universitaire de Montréal, Montreal, Quebec
  - Centre universitaire de santé McGill (CUSM), Montreal, Quebec
  - Centre Hospitalier Universitaire de Québec- Université Laval, Québec, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec (IUCPQ), Québec, Quebec
  - Centre de recherche CHUS, Sherbrooke, Quebec

REFERENCES:
- [Derived] D'Aragon F, Selzner M, Breau R, Masse MH, Lamontagne F, Masse M, Chasse M, Carrier FM, Cardinal H, Chaudhury P, Weiss M, Lauzier F, Turgeon AF, Frenette AJ, Bolduc B, Ducharme A, Lamarche C, Couture E, Holdsworth S, Bertholz L, Talbot H, Slessarev M, Luke P, Boyd JG, Shamseddin MK, Burns KEA, Zaltzman J, English S, Knoll G, Dhanani S, Healey A, Hanna S, Rochwerg B, Oczkowski SJW, Treleaven D, Meade M; Canadian Critical Care Trials Group and the Canadian Donation and Transplant Research Program. Calcineurin Inhibitor in NEuRoloGically deceased donors to decrease kidney delayed graft function study: study protocol of the CINERGY Pilot randomised controlled trial. BMJ Open. 2024 Jun 13;14(6):e086777. doi: 10.1136/bmjopen-2024-086777. PMID 38871657